CLINICAL TRIAL: NCT01624649
Title: Prospective Follow-Up Observational Study to Examine the Progression of ADHD Drug Treatment and to Analyze Associated Factors
Brief Title: A Study to Examine the Progression of Attention-Deficit Hyperactivity Disorder (ADHD) Drug Treatment and to Analyze Associated Factors
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100744; CONCERTAATT4107 (Other: Janssen Korea, Ltd., Korea); CON-KOR-5026 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Attention-deficit Hyperactivity Disorder
Keywords: Attention-deficit hyperactivity disorder; Developmental disorder; Atomoxetine; Methylphenidate; Psychiatric disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Developmental Disabilities; Mental Disorders | interventions — Methylphenidate; Atomoxetine Hydrochloride

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with ADHD: Patients will receive methylphenidate hydrochloride or atomoxetine. The methylphenidate hydrochloride is available in three forms. 1) Immediate release 2) Extended release 3) Osmotic release oral system
  Interventions: Drug: Methylphenidate hydrochloride; Drug: Atomoxetine

INTERVENTIONS:
Drug: Methylphenidate hydrochloride — Form = tablet, route = oral, administered as a flexible dosage
Drug: Atomoxetine — Form = tablet, route = oral;

SUMMARY:
The purpose of this observational study is to explore the efficacy of methylphenidate hydrochloride in children and adolescents diagnosed with attention-deficit hyperactivity disorder (ADHD) by Kiddie-scheduled for affective disorders (SADS)-present and life time version (K-SADS-PL).

DETAILED DESCRIPTION:
This is a 1-year open-label (all people involved know the identity of the assigned drug), multicenter, single arm, prospective, observational study to explore under natural setting the efficacy of drug treatment in children and adolescents diagnosed with ADHD by K-SADS-PL (K-SADS-PL is a tool used for ADHD diagnosis. Patient may be diagnosed with ADHD by using K-SADS-PL to check if he or she meets the criteria according to Diagnostic and Statistical Manual of Mental Disorders & edition (DSM-IV). After obtaining informed consent, investigator will prescribe stimulant or non-stimulant ADHD treatment medications (ie, Immediate release [IR]/extended release [ER]/osmotic release oral system (OROS) methylphenidate, atomoxetine). Efficacy and safety assessments will be performed at 4, 12, 24, 36, and 52 weeks after the first day of giving study drug. Progression of symptom improvement and adherence will be investigated and associated variables (ie, demographic, clinical, familial and treatment factors) will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Has been diagnosed with attention-deficit hyperactivity disorder (ADHD) by Kiddie-SADS-present and life time version (K-SADS-PL)
* Have not received methylphenidate or atomoxetine within 3 months prior to screening.

Exclusion Criteria:

* Has intelligence quotient (IQ) ≤70 assessed by comprehensive attention test (CAT) at screening diagnosed with congenital disorders
* Has had history of acquired brain damage (eg, cerebral palsy)
* Has had diagnosed with convulsive disabilities or other neurological disease or dysesthesia
* Has had developmental disabilities such as autistic spectrum disorder
* Has had history of schizophrenia, bipolar, or other pediatric psychotic disorder, and obsessive compulsive disorder
* Has had linguistic disability and had diagnosed with tic disorder that requires additional drug treatment.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents of age between 6 and 15 years (in Korean age) who are dianosed with ADHD by K-SADS-PL but have never received any of methylphenidate or atomoxetine within 3 months prior to screening.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the ADHD Rating Scale (ARS) | Baseline and Week 52
  The ADHD Rating Scale (ARS) - Parent Version: ARS contains 18 items, in which parent version of the questionnaire is based on home behaviors.

SECONDARY OUTCOMES:
Clinical Global Impression-Severity (CGI-S) | Baseline to Week 52
  CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Ratings are 1 = normal/not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = extremely ill.
Adherence Rate | Week 4 to Week 52
  Pill count at each visit; at least 50% adherence rate will be considered clinically relevant.
Comprehensive Attention Test (CAT) | Baseline, Week 24 and Week 52
  CAT is a computerized test which includes attention task, sustained attention to response, flanker task, divided attention task, and spatial working memory task.
Academic Performance Rating Scale (APRS) | Baseline, Week 24 and Week 52
  APRS is a 19-item scale, where parents rate the child's academic abilities and behaviors on a 5-point scale. Higher scores indicate greater academic performance.
Symptoms Checklist (SCL-90) for Parent Depression | Baseline, Week 24 and Week 52
Clinical Global Impression- Improvement (CGI-I) | Baseline and Week 52
  CGI-I is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. It is rated as 1, every much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Principal Investigator — Janssen Korea, Ltd., Korea
Locations (9):
- South Korea (9):
  - Bucheon-Si Gyeonggi-Do
  - Daegu
  - Gyeongsangnam-Do
  - Jeju Special Self-Governing Province
  - Jeonju
  - Kyunggi-Do
  - Seongnam
  - Seoul
  - Suwon